CLINICAL TRIAL: NCT05454540
Title: A Randomized Double-blinded Sham-controlled Trial of Precuneus RTMS in Mild to Moderate Alzheimer's Disease Patients.
Brief Title: Repetitive TMS of the Posterior DMN in AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Brightfocus: A2019523S
Record Dates: First submitted 2022-06-16; First posted 2022-07-12 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRANSCRANIAL MAGNETIC STIMULATION (Active Comparator): repetitive TRANSCRANIAL MAGNETIC STIMULATION (rTMS) will be applied over the precuneus. The rTMS treatment will consist of two phases: an intensive phase and a maintenance phase. The intensive phase will involve 2 weeks of treatment, 5 days per week (10 sessions, 1.600 pulses per day at 20 Hz for a total of 16.000 pulses). The maintenance phase will consist of 1 session of treatment every week for 50 weeks (80.000 pulses)
  Interventions: Device: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION
- SHAM TRANSCRANIAL MAGNETIC STIMULATION (Sham Comparator): SHAM TMS will be applied over the precuneus. The sham rTMS treatment will consist of two phases: an intensive phase and a maintenance phase. The intensive phase will involve 2 weeks of treatment, 5 days per week (10 sessions, 1.600 pulses per day at 20 Hz for a total of 16.000 pulses). The maintenance phase will consist of 1 session of treatment every week for 50 weeks (80.000 pulses)
  Interventions: Device: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION

INTERVENTIONS:
Device: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION — daily treatment session of REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION will be applied over precuneus for 20 minutes of consecutive blocks of 20Hz pulses for two seconds followed by 28 seconds of no stimulation.
  Other Name: RTMS

SUMMARY:
The primary aim of this project is to investigate the safety and efficacy of repetitive transcranial magnetic stimulation (rTMS) on cognition in patients with mild to moderate Alzheimer's disease. rTMS is considered a safe, well tolerated and relatively cheap treatment. The appealing idea of the intervention is to improve memory by directly modulating the activity of precuneus, key area linked to memory impairment. Patients will be treated with rTMS in two phases: a 2-week intensive phase followed by a maintenance phase for a total of 52 weeks. This project aims to provide a valid treatment to slow the worsening of symptoms and improve quality of life for those with Alzheimer's and their caregivers.

DETAILED DESCRIPTION:
Detailed Description:

Background: Alzheimer's disease (AD) is a neurodegenerative disorder characterized by severe disruption of large-scale brain networks connectivity. AD pathophysiology has been mainly associated with a breakdown of the Default Mode Network (DMN) and with a structural disconnection of parietal nodes. It has been shown that the precuneus (PC), a central hub of the DMN, is involved in successful episodic memory retrieval, working as a key area of the network activated by recognition memory. Recent anatomical works have shown that medial parietal regions are interconnected with the medial temporal region, which is implicated in memory retrieval. In particular, the PC was identified as a region demonstrating strong functional interconnectivity with the hippocampal formation. This is of particular relevance because PC is altered in AD. At early clinical stages of AD, PC is selectively vulnerable to early amyloid deposition, and plays a critical role in the conversion towards dementia.

Hypothesis: a novel therapeutic intervention for AD is repetitive Transcranial Magnetic Stimulation (rTMS). rTMS is a non- invasive approach that can be used to induce long lasting modulation of specific brain functions, inducing neuroplastic changes not only in the cortical site of stimulation, but also in remote interconnected areas. In a recent double blind randomized cross-over clinical pilot study, the investigators found that a two-week course of daily high-frequency rTMS (20 Hz) treatment targeting the DMN (Stimulation site: PC) was able to induce an improvement in episodic memory compared to placebo. Indeed, TMS-EEG measurements showed that rTMS treatment, applied over the DMN, was capable to modulate the cortical activity in both the targeted areas (PC) as well as in functional connected regions of the DMN.

Specific aims: to investigate clinical efficacy and safety of DMN rTMS applied during 12 months in mild to moderate AD patients. To provide novel evidence that non-invasive treatment of network dysfunction, through stimulation of the PC, will represent an effective strategy to enhance cognitive functions and lead to substantial slowing of cognitive and functional decline in patients with mild AD. The findings yielded by the present project will have a potential strong impact on clinical practice of AD patients. Since rTMS is well tolerated and relatively low-priced, a positive result could lead to a fast application of the present proposal to the clinical experience. If successful, the proposed project will provide support for a novel treatment for cognitive dysfunction in AD patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient and the responsible caregiver have signed the Informed Consent Form.
2. The patient has probable AD, diagnosed according to NINCDS-ADRDA criteria.
3. The patient is a man or woman, aged ≤ 85 years.
4. The patient has a CDR total score of 0.5 or 1 (mild to moderate) and MMSE score of 18-26 (inclusive) at Screening.
5. Has at least one identified adult caregiver
6. The patient has been treated with acetylcholinesterase inhibitor (AChEI), i.e., donepezil, galantamine, or rivastigmine, at the time of Screening

   * for at least 3 months
   * The current dosage regimen must have remained stable for ≥ 8 weeks
   * It must be planned that the dosage regimen will remain stable throughout participation in the study
7. The patient is able to comply with the study procedures in the view of the investigator.

Exclusion Criteria:

1. Significant neurodegenerative disorder of the central nervous system other than Alzheimer's disease
2. Significant intracranial focal or vascular pathology seen on brain MRI scan
3. History of seizure (with the exception of febrile seizures in childhood)
4. Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM IV-TR) criteria met for any of the following within specified period:

   * Major depressive disorder (current)
   * Schizophrenia (lifetime)
   * Other psychotic disorders, bipolar disorder, or substance (including alcohol) related disorders (within the past 5 years)
5. Metal implants in the head (except dental), pacemaker, cochlear implants, or any other non-removable items that are contraindications to MR imaging.
6. Treatment currently or within 3 months before Baseline with any of the following medications:

   * Typical and atypical antipsychotics (i.e. Clozapine, Olanzapine)
   * Antiepileptics drugs (i.e. Carbamazepine, Primidone, Pregabalin, Gabapentin)
   * Memantine

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical Dementia Rating scale (CDR) sum of boxes | change from baseline to Week 52
  global cognition and disease severity. The score range from 0-18 with the higher score meaning greater disease severity.

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) | change from baseline to Week 52
  global cognition. The score range from 0-70 with the higher score meaning greater cognitive impairment.
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | change from baseline to Week 52
  functional activities. The score range from 0-78 with a lower score indicating more severe functional impairment.
Neuropsychiatric Inventory (NPI) | change from baseline to Week 24
  behavioural symptoms. The score range from 0-144 with the higher score meaning more severe behavioural disturbances.
Frontal Assessment Battery (FAB) | change from baseline to Week 52
  frontal lobe functions. The score range from 0-18 with the higher score meaning less frontal cognitive impairment.
Cortical activity (TMS-EEG) | change from baseline to Week 52
  neurophysiological marker

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Koch, MD, PHD, Principal Investigator — Fondazione Santa Lucia IRCCS
Locations (2):
- Italy (2):
  - Giacomo Koch, Rome, <None>
  - Santa Lucia Foundation, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koch G, Casula EP, Bonni S, Borghi I, Assogna M, Di Lorenzo F, Esposito R, Maiella M, D'Acunto A, Ferraresi M, Mencarelli L, Pezzopane V, Motta C, Santarnecchi E, Bozzali M, Martorana A. Effects of 52 weeks of precuneus rTMS in Alzheimer's disease patients: a randomized trial. Alzheimers Res Ther. 2025 Apr 2;17(1):69. doi: 10.1186/s13195-025-01709-7. PMID 40176122